CLINICAL TRIAL: NCT00243230
Title: Vicriviroc (SCH 417690) in Combination Treatment With Optimized ART Regimen in Experienced Subjects (VICTOR-E1)
Brief Title: Vicriviroc (SCH 417690) in Combination Treatment With Optimized ART Regimen in Experienced Participants (VICTOR-E1) (MK-7690-020/P03672)
Acronym: VICTOR-E1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03672; 2005-001057-21 (EudraCT Number); MK-7690-020 (Other: Merck Protocol Number); P03672 (Other: Schering Corporation Protocol Number)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — vicriviroc

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There were Double-blind and an Open Label extension period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-Blind - Vicriviroc 30 mg (Experimental): Vicriviroc 30 mg once daily (QD), orally (PO), plus an open-label optimized antiretroviral therapy (ART) regimen containing a ritonavir-boosted protease inhibitor (PI/r) for 48 weeks.
  Interventions: Drug: Vicriviroc 30 mg; Drug: Background ART Regimen
- Double-Blind - Vicriviroc 20 mg (Experimental): Vicriviroc 20 mg QD, PO, plus an open-label optimized ART regimen containing a PI/r for 48 weeks.
  Interventions: Drug: Vicriviroc 20 mg; Drug: Placebo; Drug: Background ART Regimen
- Double-Blind - Placebo (Placebo Comparator): Placebo QD, PO, plus an open-label optimized ART regimen containing a PI/r for 48 weeks.
  Interventions: Drug: Placebo; Drug: Background ART Regimen
- Open-label - Vicriviroc 30 mg (Experimental): Vicriviroc 30 mg once daily (QD), orally (PO), plus an open-label optimized ART regimen containing a ritonavir-boosted protease inhibitor (PI/r) for up to 45 months.
  Interventions: Drug: Vicriviroc 30 mg; Drug: Background ART Regimen

INTERVENTIONS:
Drug: Vicriviroc 30 mg — Three tablets of vicriviroc 10 mg once daily for 48 weeks (Double-blind Period) or for up to 45 months (Open Label Period).
  Other Names: SCH 417690
  Arms: Double-Blind - Vicriviroc 30 mg; Open-label - Vicriviroc 30 mg
Drug: Vicriviroc 20 mg — Two tablets of vicriviroc 10 mg once daily for 48 weeks.
  Other Names: SCH 417690
  Arms: Double-Blind - Vicriviroc 20 mg
Drug: Placebo — Three tablets of placebo once daily for 48 weeks.
  Arms: Double-Blind - Placebo
Drug: Placebo — Two tablets of placebo once daily for 48 weeks.
  Arms: Double-Blind - Vicriviroc 20 mg
Drug: Background ART Regimen — An open-label ritonavir-boosted optimized background ART regimen containing ≥3 drugs (including a protease inhibitor [PI]) selected for each individual study participant by the investigator. The optimized regimens most commonly include new nucleoside analogs (NRTIs) and a PI, usually "boosted" with concomitant ritonavir.

SUMMARY:
Vicriviroc (vye-kri-VYE-rock) is an investigational drug that belongs to a new class of drugs, called C-C chemokine receptor type 5 (CCR5) receptor blockers. This group of drugs blocks one of the ways human immunodeficiency virus (HIV) enters T-cells (the cells that fight infection). The purpose of this 48-week study is to evaluate 2 dose levels of vicriviroc in participants with HIV who have not responded adequately to standard HIV treatments. This study was designed to evaluate the safety and efficacy of doses of vicriviroc, when taken in combination with other HIV drugs, in terms of ability to decrease the level of HIV (viral load) in the blood. The primary objective of the study was to evaluate antiviral efficacy of two doses of Vicriviroc maleate compared to placebo in combination with a protease inhibitor (PI)-containing optimized antiretroviral therapy (ART) regimen in CCR5-tropic HIV infected individuals failing a standard ART regimen.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, parallel-group, multi-center study of vicriviroc maleate in participants with HIV infected with CCR5-tropic virus only for whom standard antiretroviral treatment (ART) has failed. The study will evaluate the antiviral efficacy of two doses of vicriviroc (20 mg once daily (QD) and 30 mg QD) compared with placebo when added to optimized ART therapy. The optimized background regimen will be chosen by the investigator based on results of drug susceptibility tests, history of prior antiretroviral drug use by the participant, and drug toxicity. The background regimen must include at least 3 antiretroviral drugs (not including study drug), one of which must be a ritonavir-boosted protease inhibitor (≥100 mg ritonavir). There will be two interim analyses: when all participants have completed 12 weeks and 24 weeks of treatment, respectively. Based on the balance of safety and efficacy determined in these analyses, a dosage or dosages will be selected for further study in additional registrational trials. The primary efficacy analysis will be conducted when all participants have completed 48 weeks of treatment. After Week 48, participants who meet applicable criteria will be offered open label vicriviroc 30 mg QD, if appropriate, until the sponsor terminates the clinical development of vicriviroc. Additionally, participants who discontinue early from the study prior to Week 48 will be offered re-screening for the open label segment of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with documented HIV infection with no detectable C-X-C Motif Chemokine Receptor 4 (CXCR4)
* Prior therapy for ≥3 months with ≥3 classes of currently marketed (US FDA-approved) antiretroviral agents (nucleoside reverse transcriptase inhibitor, NRTIs, non-nucleoside reverse transcriptase inhibitor (NNRTIs), protease inhibitor (PIs), or fusion inhibitors) at any time prior to screening
* HIV ribonucleic acid (RNA) ≥1000 copies/mL on a stable ART regimen for ≥6 weeks prior to Screening and ≥8 weeks prior to randomization
* ≥1 genotypically documented resistance mutation to a reverse transcriptase (RT) inhibitor and ≥1 primary resistance mutation to a PI
* Acceptable hematologic, renal and hepatic laboratory parameters

Exclusion Criteria:

* No history of previous malignancy (with the exceptions of cutaneous Kaposi's Sarcoma without visceral or mucosal involvement that resolved with highly active antiretroviral therapy (HAART) but without systemic anti-cancer treatment, and basal-cell carcinoma of skin surgically resected with disease-free margins on pathology exam)
* Treatment with cytotoxic cancer chemotherapy,
* Recurrent seizure, or central nervous system (CNS) condition or drug use predisposing to seizure in the opinion of the investigator
* No active acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2005-09-19 (Actual); Primary Completion 2007-10-19 (Actual); Study Completion 2011-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Suleiman J, Zingman BS, Diaz RS, Madruga JV, DeJesus E, Slim J, Mak C, Lee E, McCarthy MC, Dunkle LM, Walmsley S. Vicriviroc in combination therapy with an optimized regimen for treatment-experienced subjects: 48-week results of the VICTOR-E1 phase 2 trial. J Infect Dis. 2010 Feb 15;201(4):590-9. doi: 10.1086/650342. PMID 20064072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After completing 48 weeks of blinded treatment, participants were offered open-label VCV 30 mg QD in addition to optimized background therapy (OBT). Participants who discontinued before Week 48 of the double-blind segment of the trial for reasons other than adverse events were offered rescreening for the open label extension.
Groups:
- Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen: Vicriviroc 30 mg once daily (QD), orally (PO), plus an open-label optimized antiretroviral therapy (ART) regimen containing a ritonavir-boosted protease inhibitor (PI/r) for 48 weeks.
- Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen: Vicriviroc 20 mg QD, PO, plus an open-label optimized ART regimen containing a PI/r for 48 weeks.
- Double-Blind Period - Placebo Plus an ART Regimen: Placebo QD, PO, plus an open-label optimized ART regimen containing a PI/r for 48 weeks.
- Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen: Vicriviroc 30 mg once daily (QD), orally (PO), plus an open-label optimized ART regimen containing a ritonavir-boosted protease inhibitor (PI/r) for up to 45 months.
Period: Double-Blind Period
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen
Started | 39 | 40 | 37 | 0
Treated | 39 | 40 | 35 | 0
Completed | 33 | 35 | 18 | 0
Not Completed | 6 | 5 | 19 | 0
Not completed — Adverse Event | 0 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Randomized but Not Treated | 0 | 0 | 2 | 0
Not completed — Treatment Failure - Virologic Failure defined by investigator | 5 | 3 | 14 | 0
Period: Open Label Period
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen
Started | 0 | 0 | 0 | 85
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 85
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Treatment Failure - Virologic Failure | 0 | 0 | 0 | 13
Not completed — Progressive Disease (AIDS-Event) | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Administrative Reason | 0 | 0 | 0 | 63

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen | Total
Number analyzed (Participants) | 39 | 40 | 37 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (7.3) | 44.0 (8.0) | 45.5 (8.8) | 44.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 11 | 26
  Male | 33 | 31 | 26 | 90
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 32 | 21 | 79
  Black | 9 | 3 | 8 | 20
  Asian | 0 | 1 | 0 | 1
  Other | 4 | 4 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log10 Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) at Week 48 of the Double-blind Period
Description: HIV RNA was measured by AMPLICOR HIV-1 MONITOR Standard assay. For participants who had HIV RNA below the lower quantification of the Standard assay (LOQ of 400 copies/mL), the AMPLICOR HIV-1.5 UltraSensitive assay was performed. If the HIV RNA measurement was below the lower quantification of the UltraSensitive assay (LOQ of 50 copies/mL), a value of 49 was imputed. If a continuing participant has a missing HIV RNA value at the time point of interest, the geometric mean of immediately preceding and following values was used. If the participants had no subsequent following value or discontinued study treatment before the time point of interest, then the change from baseline was set to zero. Analysis was performed with a variance (ANOVA) model that adjusted for the treatment and stratification factors (intended enfuvirtide (T20) use in current newly-optimized background regimen (OBT) (Y/N) and HIV RNA at Screening (> or ≤100,000 copies/mL)).
Time Frame: Baseline and Week 48 of the Double-blind Period
Population: The analysis population included all randomized participants who received at least 1 dose of study medication during the Double-blind Period. Participants enrolled in the Open Label Period were not included in this analysis population.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Log10 copies/mL
  Log10 HIV RNA at Baseline. | 4.52 (0.88) | 4.50 (0.89) | 4.62 (0.79)
  Change from Baseline in Log10 HIV RNA at Week 48. | -1.78 (1.31) | -1.73 (1.31) | -0.80 (1.31)
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0017, ANOVA; ANOVA model adjusted for treatment and stratification factors - the use of T20 in current OBT and the baseline HIV-1 RNA ≤100,000 copies/mL; VCV 30 mg vs. Placebo = -0.98, 95% CI 2-sided [-1.58 to -0.37]
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0026, ANOVA; [statistical method as in outcome 1, analysis 1]; VCV 20 mg vs. Placebo = -0.93, 95% CI [-1.54 to -0.33]

2. Secondary Outcome: Participants With ≥1.0 log10 Change From Baseline HIV RNA at Week 48 of the Double-blind Period
Description: HIV RNA was measured by AMPLICOR HIV-1 MONITOR Standard assay. For participants who had HIV RNA below the lower quantification of the Standard assay (LOQ of 400 copies/mL), the AMPLICOR HIV-1.5 UltraSensitive assay was performed. If the HIV RNA measurement was below the lower quantification of the UltraSensitive assay (LOQ of 50 copies/mL), a value of 49 was imputed. If a continuing participant has a missing HIV RNA value at the time point of interest, the geometric mean of immediately preceding and following values was used. If the participants had no subsequent following value or discontinued study treatment before the time point of interest, then the change from baseline was set to zero.
Time Frame: Baseline and 48 Weeks of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 26 | 25 | 12
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0052, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0190, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA

3. Secondary Outcome: Participants With HIV RNA <400 Copies/mL at Week 48 of the Double-blind Period
Description: HIV RNA was measured by AMPLICOR HIV-1 MONITOR Standard assay. For participants who had HIV RNA below the lower quantification of the Standard assay (LOQ of 400 copies/mL), the AMPLICOR HIV-1.5 UltraSensitive assay was performed. If a continuing participant has a missing HIV RNA value at the time point of interest, the geometric mean of immediately preceding and following values was used. If the participants had no subsequent following value or discontinued study treatment before the time point of interest, then the change from baseline was set to zero.
Time Frame: Week 48 of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 25 | 24 | 9
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0028, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA

4. Secondary Outcome: Participants With a Time to Loss of Virologic Response (TLOVR) Based on 0.5 Log10 Reduction by 48 Weeks of the Double-blind Period
Description: TLOVR defined as the time from randomization to either: 1. Failure to experience HIV RNA decline of ≥0.5 log10 from Baseline at Week 4, in which case time was set to 0; or 2. Rebound of HIV RNA to within 0.5 log10 of baseline value at any time after maximum suppression. HIV RNA was measured by AMPLICOR HIV-1 MONITOR Standard assay. For participants who had HIV RNA below the lower quantification of the Standard assay (LOQ of 400 c/mL), the AMPLICOR HIV-1.5 UltraSensitive assay was performed. If the HIV RNA measurement was below the lower quantification of the UltraSensitive assay (LOQ of 50 c/mL), a value of 49 was imputed. If a continuing participant has a missing HIV RNA value at the time point of interest, the geometric mean of immediately preceding and following values was used. If the participants had no subsequent following value or discontinued study treatment before the time point of interest, then the change from baseline was set to zero.
Time Frame: Up to 48 weeks of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants
  Participants with Sustained ≥0.5 Log10 Reduction by Week 4 | 31 | 32 | 15
  Participants with Rebound by Week 12 | 1 | 1 | 1
  Participants with Rebound by Week 24 | 2 | 1 | 1
  Participants with Rebound after Week 24 | 1 | 1 | 1
  Participants Suppressed through Week 48 | 27 | 29 | 12
  Participants with No ≥0.5 Log10 Reduction by Week 4 | 1 | 2 | 3

5. Secondary Outcome: Change From Baseline in Log10 HIV RNA at Week 12 of the Double-blind Period
Description: HIV RNA was measured by AMPLICOR HIV-1 MONITOR Standard assay. For participants who had HIV RNA below the lower quantification of the Standard assay (LOQ of 400 c/mL), the AMPLICOR HIV-1.5 UltraSensitive assay was performed. If the HIV RNA measurement was below the lower quantification of the UltraSensitive assay (LOQ of 50 c/mL), a value of 49 was imputed. If a continuing participant has a missing HIV RNA value at the time point of interest, the geometric mean of immediately preceding and following values was used. Missing values of change from baseline were imputed by the average of immediately preceding and following non-missing values, and in any other cases, missing values were imputed by zero.
Time Frame: Baseline and Week 12 of the Double-blind Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Log10 copies/mL
  Log10 HIV RNA at Baseline. | 4.52 (0.88) | 4.50 (0.89) | 4.62 (0.79)
  Change from Baseline in Log10 HIV RNA at Week 12. | -2.11 (1.14) | -1.94 (1.14) | -1.11 (1.14)
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0002, ANOVA; [statistical method as in outcome 1, analysis 1]; Vicriviroc 30mg - Placebo = -1.00, 95% CI 2-sided [-1.53 to -0.48]
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0020, ANOVA; [statistical method as in outcome 1, analysis 1]; Vicriviroc 20 mg - Placebo = -0.84, 95% CI 2-sided [-1.36 to -0.31]

6. Secondary Outcome: Change From Baseline in Log10 HIV RNA at Week 24 of the Double-blind Period
Description: as for outcome 5
Time Frame: Baseline and Week 24 of the Double-blind Period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Log10 copies/mL
  Log10 HIV RNA at Baseline. | 4.52 (0.88) | 4.50 (0.89) | 4.62 (0.79)
  Change from Baseline in Log10 HIV RNA at Week 24. | -2.07 (1.28) | -2.04 (1.28) | -0.96 (1.28)
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0003, ANOVA; ANOVA model adjusted for treatment and stratification factors - the use of T20 in current OBT and the baseline HIV-1 RNA <=100,000 copies/mL; Vicriviroc 30 mg - Placebo = -1.10, 95% CI 2-sided [-1.69 to -0.51]
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0004, ANOVA; [statistical method as in outcome 6, analysis 1]; Vicriviroc 20 mg - Placebo = -1.07, 95% CI 2-sided [-1.66 to -0.49]

7. Secondary Outcome: Change From Baseline CD4 Cells Count at Week 12 of the Double-blind Period
Description: Blood was collected and CD4+ cell count assessment was done by flow cytometry. Mean change from baseline in CD4 cell counts was determined. Any missing value was replaced by carrying forward baseline except if the immediately preceding and following value are available, in which case the arithmetic average of the two was used. If more than 1 CD4 count was available during a visit window, the value that was the closest to the time point of interest was used. If more than 1 pre-treatment CD4 value was available at baseline, the arithmetic mean of the 2 CD4 counts was taken.
Time Frame: Baseline and Week 12 of the Double-blind Period
Population: The analysis population included all randomized participants who received at least 1 dose of study medication and had baseline and Week 12 endpoint measurements during the Double-blind Period. Participants enrolled in the Open Label Period were not included in this analysis population.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 39 | 35
Cells/mm^3
  CD4 Cells Count at Baseline | 202.23 (159.22) | 202.10 (144.47) | 214.41 (185.62)
  Change from Baseline CD4 Cells Count at Week 12 | 109.85 (110.23) | 94.46 (110.31) | 52.09 (110.21)
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0264, ANOVA; [statistical method as in outcome 1, analysis 1]; VCV 30 mg - Placebo = 57.76, 95% CI 2-sided [6.90 to 108.61]
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.1020, ANOVA; [statistical method as in outcome 1, analysis 1]; VCV 20 mg - Placebo = 42.36, 95% CI 2-sided [-8.55 to 93.28]

8. Secondary Outcome: Change From Baseline CD4 Count at Week 24 of the Double-blind Period
Description: as for outcome 7
Time Frame: Baseline and Week 24 of the Double-blind Period
Population: The analysis population included all randomized participants who received at least 1 dose of study medication and had baseline and Week 24 endpoint measurements during the Double-blind Period. Participants enrolled in the Open Label Period were not included in this analysis population.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 39 | 35
Cells/mm^3
  CD4 Count at Baseline. | 202.23 (159.22) | 202.10 (144.47) | 214.41 (185.62)
  Change from Baseline CD4 Count at Week 24. | 97.58 (113.66) | 103.58 (113.74) | 59.46 (113.64)
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.1525, ANOVA; [statistical method as in outcome 1, analysis 1]; VCV 30 mg - Placebo = 38.12, 95% CI 2-sided [-14.32 to 90.56]
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0987, ANOVA; [statistical method as in outcome 1, analysis 1]; VCV 20 mg - Placebo = 44.12, 95% CI 2-sided [-8.38 to 96.61]

9. Secondary Outcome: Change From Baseline CD4 Count at Week 48 of the Double-blind Period
Description: as for outcome 7
Time Frame: Baseline and Week 48 of the Double-blind Period
Population: The analysis population included all randomized participants who received at least 1 dose of study medication and had baseline and Week 48 endpoint measurements during the Double-blind Period. Participants enrolled in the Open Label Period were not included in this analysis population.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 39 | 35
Cells/mm^3
  CD4 Count at Baseline. | 202.23 (159.22) | 202.10 (144.47) | 214.41 (185.62)
  Change from Baseline CD4 Count at Week 48. | 102.12 (141.68) | 133.88 (141.79) | 64.80 (141.65)
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.2603, ANOVA; [statistical method as in outcome 1, analysis 1]; VCV 30 mg - Placebo = 37.32, 95% CI 2-sided [-28.05 to 102.68]
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0387, ANOVA; [statistical method as in outcome 1, analysis 1]; VCV 20 mg - Placebo = 69.08, 95% CI 2-sided [3.64 to 134.52]

10. Secondary Outcome: Change From Baseline CD4 Count at Month 42 of the Open Label Extension
Description: Blood was collected and CD4+ cell count assessment was done by flow cytometry. Mean change from baseline in CD4 cell counts was determined. Any missing value was replaced by carrying forward baseline except if the immediately preceding and following value are available, in which case the arithmetic average of the two was used. If more than 1 CD4 count was available during a visit window, the value that was the closest to the time point of interest was used. If more than 1 pre-treatment CD4 value was available at baseline, the arithmetic mean of the 2 CD4 counts was taken. After completion of the Double-Blind Period, eligible participants could enroll in the Open Label Period and continue treatment.
Time Frame: Baseline and Month 42 of the Open Label Period
Population: The analysis population included all randomized participants who received at least 1 dose of study medication and had baseline and Month 42 endpoint measurements during the Open Label Period. Participants enrolled in the Double-blind Period were not included in this analysis population.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen
Number analyzed (Participants) | 85
Cells/mm^3
  CD4 Count at Baseline (Open Label Extension). | 366.16 (191.86)
  Change from Baseline CD4 Count at Month 42. | -78.67 (283.28)

11. Secondary Outcome: Participants With <400 Copies/mL HIV RNA at Week 12 of the Double-blind Period
Description: HIV RNA was measured by AMPLICOR HIV-1 MONITOR Standard assay. For participants who had HIV RNA below the lower quantification of the Standard assay (LOQ of 400 copies/mL), the AMPLICOR HIV-1.5 UltraSensitive assay was performed. If a continuing participant has a missing HIV RNA value at the time point of interest, the geometric mean of immediately preceding and following values was used. If the participants had no subsequent following value or discontinued study treatment before the time point of interest, then the change from baseline was set to zero. HIV RNA <400 copies/mL is a less stringent measure of viral suppression and indicates that a participant responded to treatment.
Time Frame: Week 12 of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 28 | 25 | 14
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0031, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0480, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA

12. Secondary Outcome: Participants With <400 Copies/mL HIV RNA at Week 24 of the Double-blind Period
Description: as for outcome 11
Time Frame: Week 24 of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 28 | 29 | 12
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA

13. Secondary Outcome: Number of Participants With <50, 50 to <400, and ≥400 Copies/mL HIV RNA of the Open Label Extension
Description: HIV RNA was measured by AMPLICOR HIV-1 MONITOR Standard assay (the lower quantification, [LOQ of 400 copies/mL]) and for HIV RNA below the LOQ, with the AMPLICOR HIV-1.5 UltraSensitive assay. HIV RNA <400 copies/mL is a less stringent measure of viral suppression (participant responded to treatment). HIV RNA < 50 copies/mL is a very stringent measure of viral suppression (participant achieved full virologic suppression). If a continuing participant has a missing HIV RNA value at the time point of interest, the geometric mean of immediately preceding and following values was used. Missing value for any reason will be imputed as non-responder except if the immediately preceding and following viral counts are both <50 copies/mL. Results are shown for Group 1. for participants with baseline HIV RNA <50 copies/mL, Group 2. baseline HIV RNA 50 to <400 copies/mL, and Group 3. baseline HIV RNA>400 copies/mL.
Time Frame: Up to 45 months of the Open Label Extension
Population: The analysis population included all randomized participants who received at least 1 dose of study medication during the Open Label Period. Participants enrolled in the Double-blind Period were not included in this analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen
Number analyzed (Participants) | 85
Participants
  Group 1. Baseline for RNA <50 copies/mL | 48
  Group 1. Last RNA <50 copies/mL: number analyzed (Participants) | 48
  Group 1. Last RNA <50 copies/mL | 42
  Group 1. Last RNA 50 to <400 copies/mL: number analyzed (Participants) | 48
  Group 1. Last RNA 50 to <400 copies/mL | 5
  Group 1. Last RNA ≥400 copies/mL: number analyzed (Participants) | 48
  Group 1. Last RNA ≥400 copies/mL | 1
  Group 2. Baseline for RNA 50 to <400 copies/mL | 10
  Group 2. Last RNA <50 copies/mL: number analyzed (Participants) | 10
  Group 2. Last RNA <50 copies/mL | 5
  Group 2. Last RNA 50 to <400 copies/mL: number analyzed (Participants) | 10
  Group 2. Last RNA 50 to <400 copies/mL | 2
  Group 2. Last RNA ≥400 copies/mL: number analyzed (Participants) | 10
  Group 2. Last RNA ≥400 copies/mL | 3
  Group 3. Baseline for RNA ≥400 copies/mL | 27
  Group 3. Last RNA <50 copies/mL: number analyzed (Participants) | 27
  Group 3. Last RNA <50 copies/mL | 10
  Group 3. Last RNA 50 to <400 copies/mL: number analyzed (Participants) | 27
  Group 3. Last RNA 50 to <400 copies/mL | 0
  Group 3. Last RNA ≥400 copies/mL: number analyzed (Participants) | 27
  Group 3. Last RNA ≥400 copies/mL | 15

14. Secondary Outcome: Participants With <50 Copies/mL HIV RNA at Week 12 of the Double-blind Period
Description: The lower limit of HIV RNA <50 copies/mL was determined by the UltraSensitive assay. HIV RNA <50 copies/mL is a very stringent measure of viral suppression and indicates that a participant achieved full virologic suppression. Missing value for any reason were imputed as non-responder except if the immediately preceding and following viral counts are both <50 copies/mL.
Time Frame: Week 12 of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 18 | 17 | 8
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0225, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0582, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA

15. Secondary Outcome: Participants With <50 Copies/mL HIV RNA at Week 24 of the Double-blind Period
Description: The lower limit of HIV RNA <50 copies/mL was determined by the UltraSensitive assay. HIV RNA < 50 copies/mL is a very stringent measure of viral suppression and indicates that a participant achieved full virologic suppression. Missing value for any reason will be imputed as non-responder except if the immediately preceding and following viral counts are both <50 copies/mL.
Time Frame: Week 24 of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 25 | 23 | 9
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0038, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA

16. Secondary Outcome: Participants With <50 Copies/mL HIV RNA at Week 48 of the Double-blind Period
Description: as for outcome 14
Time Frame: Week 48 of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 22 | 21 | 5
Statistical Analysis 1: Comparison: Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA
Statistical Analysis 2: Comparison: Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen vs Double-Blind Period - Placebo Plus an ART Regimen; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Cochran-Mantel Haenszel Test adjusted for stratification factors of T20 use in current OBT and baseline HIV-1 RNA

17. Secondary Outcome: Participants With Acquired Immunodeficiency Syndrome (AIDS)-Defining Events of the Double-blind Period
Description: All potential AIDS-defining events (ADEs) identified by investigators and the sponsor were submitted with supporting clinical data to an Adjudication Committee of HIV experts. These experts did not participant in the study and reviewed the data without knowledge of treatment assignment. To be analyzed as an ADE, the event required concurrence on the diagnosis by at least two of the three Adjudication Committee members. Their review consisted of available clinical and laboratory data, including relevant radiologic, endoscopic, and pathology assessments, when applicable as well as autopsy reports and/or hospital admission and discharge summaries. An independent radiologist was called upon when necessary. Guidelines for Diagnosis of AIDS-Defining Conditions (CDC's 1993 Revised Classification System for HIV Infection and Expanded Surveillance Case Definition for AIDS Among Adolescents and Adults) was used.
Time Frame: Up to 48 weeks of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 0 | 0 | 1

18. Secondary Outcome: Participants With AIDS-defining Events of the Open Label Extension
Description: All potential AIDS-defining events (ADEs) identified by investigators and the sponsor were submitted with supporting clinical data to an Adjudication Committee of HIV experts, who did not participant in the study and reviewed the blinded data. Their review consisted of available clinical and laboratory data, including relevant radiologic, endoscopic, and pathology assessments, autopsy reports and/or hospital admission and discharge summaries. An independent radiologist was called upon when necessary. Guidelines for Diagnosis of AIDS-Defining Conditions (CDC's 1993 Revised Classification System for HIV Infection and Expanded Surveillance Case Definition for AIDS Among Adolescents and Adults) was used. To be analyzed as an ADE, the event required concurrence on the diagnosis by at least 2 of 3 Adjudication Committee members. After completion of the Double-blind Period, eligible participants could enroll in the Open Label Period and continue treatment.
Time Frame: Up to 45 months of the Open Label Extension
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen
Number analyzed (Participants) | 85
Participants | 1

19. Secondary Outcome: Time to Occurrence of an AIDS-defining Event of the Double-blind Period
Description: All potential AIDS-defining events (ADEs) identified by investigators and the sponsor were submitted with supporting clinical data to an independent and blinded Adjudication Committee of HIV experts. To be analyzed as an ADE, the event required concurrence on the diagnosis by at least 2 of the 3 Adjudication Committee members. Their review included available clinical and laboratory data, including relevant radiologic, endoscopic, and pathology assessments, when applicable as well as autopsy reports and/or hospital admission and discharge summaries. An independent radiologist was called upon when necessary. Guidelines for Diagnosis of AIDS-Defining Conditions (CDC's 1993 Revised Classification System for HIV Infection and Expanded Surveillance Case Definition for AIDS Among Adolescents and Adults) was used.
Time Frame: Up to 48 weeks of the Double-blind Period
Population: The analysis population included all randomized participants who received at least 1 dose of study medication and had an AIDS-defining Event during the Double-blind Period. Participants enrolled in the Open Label Period were not included in this analysis population.
Measure: Number; unit: Days
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 0 | 0 | 1
Days |  |  | 256

20. Secondary Outcome: Observed Minimum Serum Concentration of Vicriviroc (Cmin) of the Double-blind Period
Description: Key pharmacokinetic (PK) parameters (maximum plasma concentration [Cmax], minimum plasma concentration [Cmin], area under the plasma concentration-time curve [AUC]) were estimated using a population PK modeling approach based on a two-compartment model with first-order absorption and elimination. Cmin is a measure of the minimum amount of drug in the plasma after the dose is given. Pharmacokinetics studies were not performed with participants receiving Placebo.
Time Frame: Two blood samples 2 hours apart on Week 4, Week 12, and Week 24 of the Double-blind Period
Population: The analysis population included all randomized participants who received at least 1 dose of Vicriviroc during the Double-blind Period. Pharmacokinetics studies were not performed with participants receiving Placebo. Participants enrolled in the Open Label Period were not included in this analysis population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 0
ng/mL | 206.56 (76.82) | 156.95 (62.17) |

21. Secondary Outcome: Observed Maximum (Peak) Plasma Concentration of Vicriviroc (Cmax) of the Double-blind Period
Description: Key pharmacokinetic (PK) parameters (maximum plasma concentration [Cmax], minimum plasma concentration [Cmin], area under the plasma concentration-time curve [AUC]) were estimated using a population PK modeling approach based on a two-compartment model with first-order absorption and elimination. Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Pharmacokinetics studies were not performed with participants receiving Placebo.
Time Frame: Two blood samples 2 hours apart on Week 4, Week 12, and Week 24 of the Double-blind Period
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 0
ng/mL | 316.21 (84.41) | 229.33 (61.74) |

22. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve of Vicriviroc (AUC) of the Double-blind Period
Description: Key pharmacokinetic (PK) parameters (maximum plasma concentration [Cmax], minimum plasma concentration [Cmin], area under the plasma concentration-time curve [AUC]) were estimated using a population PK modeling approach based on a two-compartment model with first-order absorption and elimination. AUC is a measure of the mean concentration levels of drug in the plasma after the dose. Pharmacokinetics studies were not performed with participants receiving Placebo.
Time Frame: Two blood samples 2 hours apart on Week 4, Week 12, and Week 24 of the Double-blind Period
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 0
hr*ng/mL | 5795.62 (1906.59) | 4314.88 (1497.70) |

23. Secondary Outcome: Participants With Detectable Vicriviroc Resistance of the Double-blind Period
Description: Resistance testing was performed at Baseline and again at the time of virologic failure or study discontinuation using the Phenosense GT assay (Monogram Biosciences, South San Francisco, CA). This assay used a combination of genotypic and phenotypic resistance techniques to determine an overall sensitivity score (OSS). The OSS represents the total number of drugs in the optimized background regimen (OBT) to which the virus was fully susceptible. Partial sensitivity is not counted towards the OSS. VCV susceptibility testing was performed with a maximal percent inhibition (MPI) plateau value of <85% as a cutoff for resistance.
Time Frame: Up to 48 weeks of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants | 1 | 4 | 0

24. Secondary Outcome: Participants With Detectable C-X-C Chemokine Receptor Type 4 (CXCR4)-Tropic Virus of the Double-blind Period
Description: Viral tropism was determined using the Monogram Trofile assay and antiviral drug susceptibility was measured by Monogram PhenoSense GT assay, based on both genotypic and phenotypic sensitivity of HIV isolates. The lower limit of sensitivity of the Trofile assay employed in this study for detection of minor X-4 using variants was 5-10%.
Time Frame: Up to 48 weeks of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants
  Participants With detectable CV (on study drug) | 9 | 7 | 3
  Participants With detectable CV with other virologic failures | 8 | 7 | 2
  Participants With detectable CV anytime who discontinued | 4 | 3 | 2

25. Secondary Outcome: Participants With Detectable CXCR4-Tropic Virus and Immune Decline (≥50% Fall in CD4 Count From Baseline) of the Double-blind Period
Description: Viral tropism was determined using the Monogram Trofile assay and antiviral drug susceptibility was measured by Monogram PhenoSense GT assay, based on both genotypic and phenotypic sensitivity of HIV isolates. The lower limit of sensitivity of the Trofile assay employed in this study for detection of minor X-4 using variants was 5-10%. Participants with emergence of CXCR4 tropism who had a concomitant decline in CD4 count by ≥50% below baseline was also computed.
Time Frame: Up to 48 weeks of the Double-blind Period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen
Number analyzed (Participants) | 39 | 40 | 35
Participants
  Participants with detectable CXCR4 virus pretreatment | 3 | 1 | 2
  Participants with ≥50% fall in CD4 count from baseline | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 weeks for the Double-blind Period Up to 45 months for the Open Label Period.
Description: The analysis population for adverse events included all randomized participants who received at least one dose of study drug during the Double-Blind Treatment Period and during the Open Label Extension. The analysis population for All-Cause Mortality was the all randomized population. MedDRA Version 10.1 was used for analysis of the Double-Blind Treatment Period data, and Version 13.1 was used for analysis of the Open Label Extension data.
Arm/Group | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen | Double-Blind Period - Placebo Plus an ART Regimen | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen
All-Cause Mortality (participants affected / at risk) | 0/39 | 2/40 | 2/37 | 1/85
Serious Adverse Events (participants affected / at risk) | 4/39 | 5/40 | 5/35 | 13/85
Other Adverse Events (participants affected / at risk) | 34/39 | 31/40 | 29/35 | 58/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen (N=39) | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen (N=40) | Double-Blind Period - Placebo Plus an ART Regimen (N=35) | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen (N=85)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERICARDITIS URAEMIC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS ESCHERICHIA COLI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATINE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LACUNAR INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URETERIC OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETROPERITONEAL LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPLASTIC NAEVUS SYNDROME (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Urinary Tract Infection
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PENIS CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSKINESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYSTERECTOMY (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SALPINGO-OOPHORECTOMY BILATERAL (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL FUSION SURGERY (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Period - Vicriviroc 30 mg Plus an ART Regimen (N=39) | Double-Blind Period - Vicriviroc 20 mg Plus an ART Regimen (N=40) | Double-Blind Period - Placebo Plus an ART Regimen (N=35) | Open-Label Period - Vicriviroc 30 mg Plus an ART Regimen (N=85)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 3 (5) | 6 (6) | 2 (2) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 15 (17) | 11 (17) | 9 (13) | 9 (10)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 3 (5) | 5 (7) | 2 (2)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
ASTHENIA (General disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (2)
FATIGUE (General disorders) | 2 (2) | 5 (6) | 3 (3) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 2 (4) | 3 (3)
PYREXIA (General disorders) | 4 (4) | 4 (8) | 4 (5) | 6 (9)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
BRONCHITIS (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 6 (10)
FOLLICULITIS (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 8 (11)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (4)
ONYCHOMYCOSIS (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 1 (2)
ORAL CANDIDIASIS (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
SINUSITIS (Infections and infestations) | 2 (2) | 4 (5) | 2 (2) | 10 (12)
TINEA PEDIS (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 11 (15)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
LIPASE INCREASED (Investigations) | 3 (5) | 0 (0) | 2 (3) | 1 (1)
WEIGHT DECREASED (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 1 (1) | 5 (6)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (3) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 5 (7)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
DIZZINESS (Nervous system disorders) | 5 (5) | 1 (1) | 4 (5) | 1 (1)
HEADACHE (Nervous system disorders) | 5 (5) | 3 (4) | 7 (8) | 7 (10)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
DEPRESSION (Psychiatric disorders) | 3 (3) | 4 (4) | 6 (6) | 3 (3)
INSOMNIA (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2) | 5 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (7) | 2 (2) | 7 (10)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
SKIN NODULE (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 5 (6)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or for presentation, review copies of the publication or presentation for review and comment on the data analysis and presentation including proprietary information, the accuracy of the information, and to ensure compliance with FDA regulations.